CLINICAL TRIAL: NCT02340637
Title: Coping Kids: A Randomized Controlled Study of a New Indicated Preventive Intervention for Children With Symptoms of Anxiety and Depression
Brief Title: Coping Kids: Early Intervention for Anxiety and Depression
Acronym: TIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionsenter for barn og unges psykiske helse (Other)
Collaborators: The Research Council of Norway (Other); Regional kunnskapssenter for barn og unge - Midt (Unknown); Regional kunnskapssenter for barn og unge - Nord (Unknown)
Responsible Party: Principal Investigator, Simon-Peter Neumer, Senior Researcher, Regionsenter for barn og unges psykiske helse
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 228846/H10
Record Dates: First submitted 2014-06-12; First posted 2015-01-16 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coping Kids (Experimental): A Program for Managing Anxiety and Depression (P.C Kendall et al., 2013) is a newly developed group intervention targeting children aged 8 to 13 years who experience difficulty with symptoms of anxiety, depression, or both. The program is designed as an indicated prevention intervention to reduce the symptom levels and reduce the likelihood of the development of an anxiety disorder and/or depression.
  The youth-focused sessions are designed for implementation in school settings, and the program includes parent group meetings.
  All groupleaders participate in a three days training, followed by supervision. Manuals and workbooks are provided by the project. In addition is the same presentation as in TAU offered to the schools.
  Interventions: Behavioral: Coping Kids
- TAU (Active Comparator): The teachers and school-nurses in the control schools will conduct treatment as usual (TAU).The project offers a 2,5 hours presentation to the schools, providing general information about the research study, the prevalence of emotional disorders and how to handle emotional disorders in treatment as usual. No materials are provided by the project.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Coping Kids — The first half (10 sessions) of Coping Kids focuses on building skills that are common to both anxiety and depression. The children practice strategies to regulate their mood, learn problem-solving, and behavioral activation is used to break the cycle of withdrawal. The second half of Coping Kids (10 sessions) is focused on the youth's specific problem; for depressive symptoms, building a positive self-schema and behavioral activation; for anxiety problems, gradual exposure to fear-inducing situations. Cognitive restructuring directed at different maladaptive thoughts is also emphasized.
  Other Names: TIM
  Arms: Coping Kids
Behavioral: TAU — Treatment as usual
  Arms: TAU

SUMMARY:
The purpose of this study is to provide knowledge regarding the effect of early intervention and prevention on the development of anxiety and depression in children. The focus of the intervention is to reduce symptoms of anxiety and depression and help children develop skills to enhance self-esteem in order to improve life quality. Gender and ethnicity will be studied as moderating factors. Primary care givers will be trained in the use of evidence based methods for children with internalizing difficulties. Children in need will be identified and receive improved services, based on international standards. Active collaboration will be established nationally between three Centers for child and adolescent mental health (RKBU/RBUP) and internationally with Philip C. Kendall at the Temple University in Philadelphia and Kevin Stark at University of Texas at Austin.

Primary aims are to examine if an indicated group and school based program, Coping Kids, is more effective than treatment as usual (TAU) in reducing high levels of symptoms of both anxiety and depression among 8-12 year old schoolchildren, and if the the effects are stable over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children at the intervention schools indicating a symptom level of, at minimum, one standard deviation above mean on anxiety and/or depression on self-report measures will be offered participation in an intervention group

Exclusion Criteria:

* Children who for different reasons may not benefit from a group-process intervention (e.g. mental retardation) will be considered individually and the reasons for exclusion will be documented in the Consort flow-chart.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 873 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
MASC-C (Multidimensional Anxiety Scale for Children) | baseline, 10 weeks, 12 month
  Children: (1) MASC-C (March, 1997): A 40- items self-report assessing change in anxiety in children and adolescents between 8 and 19 years.
MFQ (Mood and Feelings Questionnaire-short version) | baseline, 10 weeks, 12 months
  Children: (2) MFQ short Version (Angold et al., 1994): A 13-items measure assessing change in cognitive, affective and behavioral-related symptoms of depression in children 8 to 18 years, with one added question about suicidality.

CONTACTS AND LOCATIONS:
Overall Officials: Simon-Peter Neumer, Dr. phil, Principal Investigator — Regionsenter for barn og unge psykiske helse
Locations (3):
- Norway (3):
  - Regionsenter for barn og unges psykiske helse, Oslo
  - Regional kunnskapssenter for barn og unge - Nord, Tromsø
  - Regional kunnskapssenter for barn og unge - Midt, Trondheim

REFERENCES:
- [Result] Patras J, Martinsen KD, Holen S, Sund AM, Adolfsen F, Rasmussen LP, Neumer SP. Study protocol of an RCT of EMOTION: An indicated intervention for children with symptoms of anxiety and depression. BMC Psychol. 2016 Sep 26;4(1):48. doi: 10.1186/s40359-016-0155-y. PMID 27671742
- [Result] Martinsen KD, Neumer SP, Holen S, Waaktaar T, Sund AM, Kendall PC. Self-reported quality of life and self-esteem in sad and anxious school children. BMC Psychol. 2016 Sep 13;4(1):45. doi: 10.1186/s40359-016-0153-0. PMID 27624487
- [Derived] Pedersen ML, Jozefiak T, Sund AM, Holen S, Neumer SP, Martinsen KD, Rasmussen LMP, Patras J, Lydersen S. Psychometric properties of the Brief Problem Monitor (BPM) in children with internalizing symptoms: examining baseline data from a national randomized controlled intervention study. BMC Psychol. 2021 Nov 27;9(1):185. doi: 10.1186/s40359-021-00689-1. PMID 34838153
- [Derived] Rasmussen LP, Patras J, Handegard BH, Neumer SP, Martinsen KD, Adolfsen F, Sund AM, Martinussen M. Evaluating Delivery of a CBT-Based Group Intervention for Schoolchildren With Emotional Problems: Examining the Reliability and Applicability of a Video-Based Adherence and Competence Measure. Front Psychol. 2021 Jun 28;12:702565. doi: 10.3389/fpsyg.2021.702565. eCollection 2021. PMID 34262514
- [Derived] Martinsen KD, Rasmussen LP, Wentzel-Larsen T, Holen S, Sund AM, Pedersen ML, Lovaas MES, Patras J, Adolfsen F, Neumer SP. Change in quality of life and self-esteem in a randomized controlled CBT study for anxious and sad children: can targeting anxious and depressive symptoms improve functional domains in schoolchildren? BMC Psychol. 2021 Jan 21;9(1):8. doi: 10.1186/s40359-021-00511-y. PMID 33478593
- [Derived] Loevaas MES, Lydersen S, Sund AM, Neumer SP, Martinsen KD, Holen S, Patras J, Adolfsen F, Rasmussen LP, Reinfjell T. A 12-month follow-up of a transdiagnostic indicated prevention of internalizing symptoms in school-aged children: the results from the EMOTION study. Child Adolesc Psychiatry Ment Health. 2020 Apr 22;14:15. doi: 10.1186/s13034-020-00322-w. eCollection 2020. PMID 32336987
- [Derived] Pedersen ML, Holen S, Lydersen S, Martinsen K, Neumer SP, Adolfsen F, Sund AM. School functioning and internalizing problems in young schoolchildren. BMC Psychol. 2019 Dec 23;7(1):88. doi: 10.1186/s40359-019-0365-1. PMID 31870462